CLINICAL TRIAL: NCT02966262
Title: Optical Coherence Tomography Registry of Korea University Anam Hospital
Brief Title: Korea University Anam Hospital Optical Coherence Tomography Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Dr. Cheol Woong Yu, MD, PhD, Korea University Anam Hospital
Other Study IDs: KUMC
Record Dates: First submitted 2016-04-25; First posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Artery Disease; Optical Coherence Tomography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Optical Coherence Tomography registry group: Patients who had undergone optical coherence tomography within coronary intervention
  Interventions: Device: Optical coherence tomography

INTERVENTIONS:
Device: Optical coherence tomography — Intracoronary imaging device which can precisely observe intracoronary structures

SUMMARY:
All comer registry who had undergone intravascular optical coherence tomography during and/or after coronary intervention.

DETAILED DESCRIPTION:
Optical coherence tomography registry is composed with before coronary stenting, immediate after coronary stenting and follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* patients who had undergone coronary intervention and optical coherence tomography

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All comer registry with patients who had undergone coronary intervention and optical coherence tomography
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of participants with Major Adverse Cardiovascular Events (MACE) | Up to 10 years
  Composite of non-fatal myocardial infarction, all cause death, target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Do-Sun Lim, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No